CLINICAL TRIAL: NCT05496088
Title: Persistent AF Catheter Ablation: Re-PVI Vs. Re-PVI + Continuous Complex Activity Mapping and Ablation - AF-CAM
Acronym: AF-CAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios proresearch (Industry)
Collaborators: Asklepios Klinik St. Georg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #3759
Record Dates: First submitted 2022-06-27; First posted 2022-08-11 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Ablation strategy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, open-label, blinded endpoint, multi-center study to compare the efficacy of adding additional ablation step (targeting areas of complex, continuous electrical activity in LA) beyond Re-PVI during catheter ablation of Atrial Fibrillation (AF) in patients undergoing 2nd ablation procedure.
  Trial flow Patients fitting the enrollment criteria and signing the informed consent form will be included and will undergo the Redo procedure for catheter ablation of pers. AF. After Re-PVI only patients with ongoing or inducted AF will be randomized. Patients, who do not fulfill this intraprocedural criteria for randomization will not be randomized but be treated as dropouts.
  Randomization is based on a 1:1 ratio into two study arms:
  1. RePVI only: Re-PVI (followed by cardioversion if AF persists)
  2. RePVI + substrate ablation: Re-PVI followed by ablation of areas of complex, continuous activity (followed by cardioversion if AF persists).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Re-PVI only (Active Comparator): Repeat ablation of pulmonary veins (Re-PVI), followed by electrical cardioversion if AF persists, n=100 pts
  Interventions: Procedure: Re-PVI only
- Group 2: Re-PVI + substrate ablation (Active Comparator): Repeat ablation of pulmonary veins (Re-PVI) + mapping & ablation of areas of continuous, complex activity, n=100 pts
  Interventions: Procedure: Re-PVI only; Procedure: Re-PVI + substrate ablation

INTERVENTIONS:
Procedure: Re-PVI only — Comparison of two treatment strategies of persistent AF catheter ablation:
  Re-PVI vs. Re-PVI + continuous complex activity mapping and ablation.
  Other Names: Repeat-PVI followed by electrocardioversion if AF persists
Procedure: Re-PVI + substrate ablation — Comparison of two treatment strategies of persistent AF catheter ablation:
  Re-PVI vs. Re-PVI + continuous complex activity mapping and ablation.
  Other Names: Repeat-PVI followed by mapping & ablation of areas of continuous, complex activity
  Arms: Group 2: Re-PVI + substrate ablation

SUMMARY:
Major objective is to compare the efficacy of adding additional ablation step (targeting areas of complex, continuous electrical activity in LA) beyond Re-PVI during catheter ablation of Atrial Fibrillation (AF) in patients undergoing 2nd ablation procedure.

Underlying hypothesis that in addition, to Re-PVI, an ablation step targeting areas of complex continuous activity will increase atrial arrhythmias freedom compared to Re-PVI only ablation.

DETAILED DESCRIPTION:
Catheter ablation of atrial fibrillation (AF) became first-line therapy in patients not responding to electrical or pharmacological cardioversion. In case of paroxysmal AF, pulmonary vein isolation (PVI) aiming at complete electrical isolation is recommended due to high acute and long term success rates. However, once AF becomes persistent, ablation efficiency dramatically decreases, most likely due to advanced electrical and structural remodeling of the atria.

Some studies, most notably STAR AF II and CHASE AF suggested that additional ablation beyond PVI may not benefit patients as expected. In parallel to studies questioning additional ablation, several studies exploring novel promising techniques were published reporting positive results, e.g. high frequency source ablation, electrogram complexity guided ablation, low voltage amplitude, activation dispersion guided ablation, stepwise ablation approach, autonomic ganglia modification and techniques of identification of rotating waves and point sources to name just few.

Such contrasting studies left EP community confused with regards to the strength of reported claims and practical recommendations. Thus, presently, there is no standard approach to AF substrate ablation and specifics regarding targets and technique are left to physician discretion, most likely resulting in a delivery of unnecessary treatment and obstructing identification of valuable approaches. Thus, there is a need for further studies exploring additional ablation techniques in a rigorous, randomized studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent atrial fibrillation, defined as atrial fibrillation which is:

   * Sustained beyond 7 days but no more than one year.
   * Or lasting less than 7 days, but with at least one episode longer than 48 h and necessitating pharmacologic or electrical cardioversion.
2. Documentation of atrial fibrillation on either a 12-lead ECG or ambulatory holter monitoring or telemetry strip.
3. One previous PVI only procedure in 3 years previous, but not within the last 3 months.
4. Age 18 - 80 years.
5. Patient is willing to participate in the study (signed written informed consent)
6. Patient is willing and available to perform all follow ups.

Exclusion Criteria:

1. Atrial fibrillation due to reversible causes.
2. Continuous AF > 12 months.
3. Any cardiac surgery within the past 2 months (60 days).
4. Documented LA thrombus on imaging.
5. LA size >60 mm.
6. Contraindication to anticoagulation (heparin or warfarin).
7. Myocardial infarction within the past 2 months (60 days).
8. Documented thromboembolic event (including TIA) within the past 12 months.
9. Rheumatic Heart Disease.
10. Uncontrolled heart failure or NYHA function class III or IV.
11. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days).
12. Unstable angina.
13. Acute illness or active systemic infection or sepsis.
14. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
15. Diagnosed atrial myxoma.
16. Significant severe pulmonary disease, (eg, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
17. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
18. Women who are pregnant (as evidenced by pregnancy test if pre- menopausal).
19. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter.
20. Presence of a condition that precludes vascular access.
21. Patients with hemodialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia | through 3 to 12 months
  Freedom from any form of sustained atrial arrhythmia (>30 s) follow-up on either a 12 lead ECG on visits or on 48h holter monitoring or on symptom driven event monitoring

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Vivantes - Klinikum Am Urban, Berlin
  - Evangelisches Krankenhaus Duesseldorf, Düsseldorf
  - Asklepios Klinik St. Georg, Hamburg